CLINICAL TRIAL: NCT03337295
Title: The Correlation Between the Thickness of Lipid Layer and the Meibomian Gland
Brief Title: The Correlation Between the Thickness of Lipid Layer and the Meibomian Gland Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Attending Doctor, Wenzhou Medical University
Other Study IDs: MJL-WZMC
Record Dates: First submitted 2016-10-14; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian Gland Dysfunction; Lipid Layer Thickness
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Low-MGD
- High-MGD

SUMMARY:
The purpose of this study is to assess the correlation between the thickness of lipid layer and the meibomian gland dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent the Meibomian Gland Dysfunction through the signs.

Exclusion Criteria:

* Eye surgery history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was consisted of patients who underwent the Meibomian Gland Dysfunction through the signs. The Office of Research Ethics,Eye Hospital of Wenzhou Medical University approved the study protocol, and all patients provided their informed consent.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Lipid Layer Thickness | up to 2 years

SECONDARY OUTCOMES:
Atrophy of Meibomian Gland | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yun-e Zhao, MD, Study Chair — Wenzhou Medical University
Locations (1):
- Wenzhou Medical University, Wenzhou, Zhejiang, China